CLINICAL TRIAL: NCT01493817
Title: Observational - Relationships Between Tumor-Associated Macrophages and Clinicopathological Factors in Wilms Tumor
Brief Title: Biomarkers in Samples From Younger Patients With Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN12B1; NCI-2012-00093 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Wilms Tumor and Other Childhood Kidney Tumors
MeSH Terms: conditions — Wilms Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basic science (biomarker analysis): Paraffin-embedded specimens are analyzed for macrophage markers. Results of each sample are then compared with patient's tumor stage, presence of vascular invasion, tumor progression, and survival.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is studying biomarkers in tissue samples from younger patients with Wilms tumor. Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how patients respond to treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether recruitment of tumor-associated macrophages is related to clinicopathological factors in Wilms tumor (tumor stage, presence of vascular invasion, tumor progression, and survival).

OUTLINE:

Paraffin-embedded specimens are analyzed for macrophage markers. Results of each sample are then compared with patient's tumor stage, presence of vascular invasion, tumor progression, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Wilms tissue microarray samples provided by the Children's Oncology Group

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Wilms tumor patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Relationship of tumor-associated macrophages and prognosis | 1 month
  Correlation of each type of macrophage score with tumor staging, presence of vascular invasion, and disease-free survival will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kandel, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States